CLINICAL TRIAL: NCT07193836
Title: Synergistic Effect of Intravenous Lidocaine on Anesthetic Induction and Emergence in Patients Undergoing Laparoscopic Cholecystectomy or Gynecological Surgery
Acronym: Li
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Huiwen Zhang-2025-09
Record Dates: First submitted 2025-09-02; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cholecystectomy, Laparoscopic; Gynecologic Surgical Procedures; Anesthesia and Procedure Related Time Intervals
Keywords: Lidocaine; General anesthesia; Consciousness; EEG monitoring; PSi index; Anesthesia induction
MeSH Terms: interventions — Saline Solution; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study uses a quadruple-blind design. Participants, care providers, investigators, and outcome assessors were blinded to group allocation to minimize performance and assessment bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1. Placebo Group (Placebo Comparator): Participants received an intravenous injection of 0.9% normal saline at induction, with no lidocaine administration throughout the perioperative period.
  Interventions: Drug: Normal Saline (0.9% NaCl)
- 2. Lidocaine Bolus Group（Experimental） (Experimental): Participants received a single intravenous bolus of lidocaine (1.5 mg/kg) at anesthesia induction. No continuous infusion was administered.
  Interventions: Drug: Lidocaine
- 3. Lidocaine Bolus + Infusion Group（Experimental） (Experimental): Participants received an intravenous bolus of lidocaine (1.5 mg/kg) at induction, followed by continuous intravenous infusion of lidocaine (2.0 mg/kg/h) until the end of surgery.
  Interventions: Drug: Lidocaine Bolus + Infusion

INTERVENTIONS:
Drug: Normal Saline (0.9% NaCl) — Participants in the control group received a single intravenous injection of 0.9% normal saline at induction of anesthesia.
  Arms: 1. Placebo Group
Drug: Lidocaine — Participants in this group received a single intravenous bolus of lidocaine (1.5 mg/kg) at anesthesia induction. No additional lidocaine was administered thereafter.
  Arms: 2. Lidocaine Bolus Group（Experimental）
Drug: Lidocaine Bolus + Infusion — Participants in this group received a bolus of lidocaine (1.5 mg/kg) at induction followed by continuous intravenous infusion of lidocaine (2 mg/kg/h) until the end of surgery.
  Arms: 3. Lidocaine Bolus + Infusion Group（Experimental）

SUMMARY:
This study aims to evaluate the effect of intravenous lidocaine on consciousness changes during anesthesia in patients undergoing laparoscopic cholecystectomy or gynecologic surgery. A total of 150 patients will be randomly assigned to one of three groups: a single-dose lidocaine group, a continuous-infusion group, or a placebo group. All patients will receive standard anesthesia care, and the study will monitor brain activity using EEG-based PSi values to measure anesthesia induction time, recovery time, and changes in consciousness. The goal is to determine whether lidocaine can reduce the amount of anesthetic used, shorten the time to fall asleep, and promote faster awakening after surgery. The results may help improve anesthesia safety and enhance recovery in surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years.
* ASA physical status I-III.
* Scheduled for elective laparoscopic cholecystectomy, laparoscopic
* hysterectomy, or laparoscopic ovarian cystectomy.
* Expected surgical duration < 120 minutes.
* Preoperative normal cognitive function (MoCA > 26).
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Known allergy to lidocaine or other amide-type local anesthetics.
* History of severe arrhythmias, heart failure (NYHA class III or higher), or epilepsy.
* Central nervous system disorders (e.g., stroke, brain trauma, seizure disorders) or psychiatric illness.
* Severe hepatic or renal dysfunction (ALT/AST > 2× ULN, or eGFR < 60 ml/min/1.73 m²).
* Currently taking medications that affect CNS function (e.g., benzodiazepines, antidepressants, antiepileptics).
* Pregnant or breastfeeding women.
* History of drug or alcohol dependence.
* BMI > 30 kg/m² or < 18 kg/m².
* Inability to understand study procedures or refusal to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to emergence from general anesthesia | Immediately after anesthesia discontinuation (Day 0)
  Measured as the time interval (in seconds) from discontinuation of anesthetics to eye opening on verbal command.
Time to loss of consciousness | During anesthesia induction on Day 0
  Measured as the time (in seconds) from the beginning of propofol administration to loss of response to verbal command and eyelash reflex.

SECONDARY OUTCOMES:
Total propofol dosage during anesthesia induction | During anesthesia induction on Day 0
  Total amount of propofol (in mg) administered from the start of anesthesia to the achievement of loss of consciousness.
Total amount of propofol administered during the entire surgical procedure | During the surgical procedure on Day 0
  Total amount of propofol (in mg/kg/h) administered during the entire surgical procedure
Mean Arterial Pressure (MAP) | Baseline, intraoperative (Day 0), and immediately post-anesthesia (Day 0)
  MAP will be recorded at three time points: prior to induction of anesthesia (baseline), during anesthesia maintenance, and after emergence from anesthesia. Unit of Measure: mmHg
Heart Rate (HR) | Baseline, intraoperative (Day 0), and immediately post-anesthesia (Day 0)
  HR will be recorded at three time points: prior to induction of anesthesia (baseline), during anesthesia maintenance, and after emergence from anesthesia. Unit of Measure: beats per minute (bpm)
Oxygen Saturation (SpO₂) | Baseline, intraoperative (Day 0), and immediately post-anesthesia (Day 0)
  SpO₂ will be recorded at three time points: prior to induction of anesthesia (baseline), during anesthesia maintenance, and after emergence from anesthesia. Unit of Measure: %
Change in Patient State Index (PSI) values at four key timepoints | Baseline, intraoperative (Day 0), and immediately post-anesthesia (Day 0)
  PSI will be measured using the Masimo SedLine® monitor at:
  Baseline (before induction) After loss of consciousness Minimum value during anesthesia After emergence The difference in PSI between timepoints will be analyzed.

OTHER OUTCOMES:
Incidence of intraoperative hypotension or bradycardia | Intraoperative period (Day 0)
  Number of participants experiencing mean arterial pressure (MAP) <65 mmHg and/or heart rate (HR) <50 bpm requiring pharmacological intervention during surgery.
Incidence of perioperative adverse drug reactions related to propofol or lidocaine | From start of anesthesia induction to 1 hour after emergence (Day 0)
  Adverse drug reactions (ADRs) related to propofol or lidocaine administration will be monitored and recorded during the perioperative period. Specific reactions include, but are not limited to:
  * Hypotension (MAP < 65 mmHg)
  * Bradycardia (HR < 50 bpm)
  * Apnea or respiratory depression
  * Pain on injection
  * Allergic reactions (e.g., rash, pruritus)
  * Delayed emergence from anesthesia
  * Neurological symptoms (e.g., dizziness, perioral numbness)
Postoperative quality of recovery score | Within 24 hours after surgery
  Assessed using a validated quality of recovery questionnaire (e.g., QoR-15 or equivalent), evaluating domains such as physical comfort, emotional state, pain, independence, and support.
Use of doxapram during the emergence phase of anesthesia | From cessation of anesthetic agents to 30 minutes post-emergence (Day 0)
  The number of participants who receive intravenous doxapram during the emergence phase from general anesthesia will be recorded. Doxapram administration is considered if spontaneous breathing or consciousness recovery is delayed beyond clinical expectations. Time of administration, total dose, and reason for use will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No